CLINICAL TRIAL: NCT03585621
Title: A Phase I-II Study of Stereotactic Body Radiation Therapy for Breast Cancer (SBRT Breast)
Brief Title: Stereotactic Body Radiation Therapy for Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Sunnybrook Regional Cancer Centre (Other)
Responsible Party: Principal Investigator, Danny Vesprini, MD, MSc, FRCPC, Deputy Chief, Department of Radiation Oncology - Clinical Care, Toronto Sunnybrook Regional Cancer Centre
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 003-2017
Record Dates: First submitted 2018-06-19; First posted 2018-07-13 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Sequential dose escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT to the Primary Breast Tumour (Experimental): SBRT to the breast using 4 sequentially escalating dose levels from 9Gy to 12 Gy.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Each radiation treatment plan will be customized to the patient and tumour in order to deliver highly conformal, conebeam CT guided SBRT radiotherapy in 4 fractions delivered over 2-4 weeks.
  Other Names: SABR

SUMMARY:
This is a prospective, single institution, phase I-II study of stereotactic body radiotherapy (SBRT) for unresected breast cancer. Twenty-four patients with advanced breast cancer who are not candidates for surgery (metastatic disease, unresectable, medically inoperable) or decline surgery will be enrolled in a prospective study using SBRT (4 fractions of radiation therapy over 12-15 days) as the primary treatment modality.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diagnosis of invasive breast carcinoma of non-lobular histology.

Unifocal tumour Previously assessed by a breast surgeon and medical oncologist, with no surgery being recommended at time of enrollment.

Primary breast and axillary surgery not recommended/performed due to any of the following:

* distant metastatic disease
* unresectable T4 disease and/or
* medically inoperable and/or
* patient declined breast surgery Stages T1-T4, N1-N2, M0-M1 disease Ability to attend radiation planning and therapy, able to attend for follow-up care Able to provide written informed consent.

Exclusion Criteria:

Received chemotherapy within 3 weeks prior to breast SBRT. (Concurrent endocrine therapy is permitted) Multifocal or multicentric tumours. Ipsilateral supraclavicular or infraclavicular nodal disease >= 1cm size that is at the level of or superior to the brachial plexus Unable to meet the brachial plexus dose constraints despite compromising coverage of target volumes - as per the discretion of the treating physician Treatment target volume estimated to occupy > 50% of the ipsilateral whole breast volume.

Locally recurrent breast cancer, with previous radiotherapy to the breast, or previous lumpectomy or mastectomy. Ipsilateral breast implant. Serious non-malignant disease that precludes definitive surgical or radiation treatment (e.g.

scleroderma, systemic lupus erythematosus, cardiovascular/pulmonary/renal disease).

Women who are pregnant or lactating. Psychiatric or addictive disorders that preclude obtaining informed consent or adherence to protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-07-17 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 12 weeks post treatment
  Incidence of side effects /toxicity associated with SBRT to the breast, during and in the three months following treatment using CTCAE v4.0

SECONDARY OUTCOMES:
Breast Symptom Scores | 2 years post treatment
  Patient reported breast symptom scores for bleeding, discharge and odour measured on a scale from 1 (no symptoms) to 10 (worst possible/continuous symptoms) using the Visual Analogue Scale tool
Patient Reported Quality of Life | 2 years post treatment
  Patient reported quality of life measured using the combined EORTC QLQ-C30 and QLQ-BR23 questionnaires
Patient Reported Quality of Life | 2 years post treatment
  Patient reported quality of life measured using the VES13 questionnaire.
Patient Reported Pain Level | 2 years post treatment
  Patient reported pain levels measured on a scale from 1 (no pain) to 10 (maximum pain tolerable) using the Visual Analogue Scale for Pain
Tumour Response Rate | 2 years post treatment
  Measured on follow-up MRI or CT imaging using RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Danny Vesprini, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No